CLINICAL TRIAL: NCT05561348
Title: Study on the Therapeutic Effect and Brain Mechanism of Transcutaneous Vagal Nerve Stimulation on Gait Impairments in Parkinson's Disease
Brief Title: The Effect and Mechanism of Transcutaneous Auricular Vagus Nerve Stimulation on Gait Impairments in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kezhong Zhang, professor，Chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-SR-535
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
Keywords: gait; Therapeutics
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active transcutaneous auricular vagus nerve stimulation (Experimental): For Experimental Arm, active transcutaneous auricular vagus nerve stimulation, Patients underwent seven consecutive daily sessions of taVNS.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation
- sham transcutaneous auricular vagus nerve stimulation (Sham Comparator): For sham transcutaneous auricular vagus nerve stimulation arm, Sham Comparator, patients underwent seven consecutive daily sessions of sham-taVNS (the electrodes were fixed at the same position without releasing current).
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — Transcutaneous auricular vagus nerve stimulation was conducted by transcutaneous electrical stimulation therapy instrument to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs, twice a day, 30 minutes each time. In the sham stimulation group, the electrodes were fixed at the same position without releasing current.

SUMMARY:
This study is a double blind comparative study examining the effectiveness of the transcutaneous auricular vagus nerve stimulation treatment on Parkinson's disease patients . We hypothesize that treatment using transcutaneous auricular vagus nerve stimulation will improve gait impairments and cortical activity in Parkinson's disease patients.

DETAILED DESCRIPTION:
Patients in the Experimental group underwent seven consecutive daily sessions of transcutaneous auricular vagus nerve stimulation (taVNS, twice daily, 30 minutes each time) , whereas patients in the sham stimulation group underwent seven consecutive daily sessions of sham taVNS. Assessments of gait function, motor symptoms and cortical activity (using Functional near-infrared spectroscopy) were performed two times: at baseline, one day post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease (PD), as diagnosed by a neurologist.
2. Hoehn and Yahr stage ≤ 2 during ON medication state.
3. Age between 40 and 80 years old.
4. Mini-Mental State Examination score >24.
5. Ability to walk at least 60s independently.
6. Stable medication

Exclusion Criteria:

1. Patients with significant visual impairment or coexisting local or systemic diseases (e.g. osteoarthritis or other neurological conditions) likely to affect gait were excluded from our study.
2. Patients who underwent deep brain stimulation surgery or those with an implanted cardiac pacemaker were also excluded
3. Patients with known or suspected cardiovas-cular disease, uncontrolled hypertension or recent myocardial infarction were also excluded from the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Velocity at one day post intervention | Assessed at baseline, one day post intervention
  The velocity will be recorded in cm/s.
Change from Baseline Step length at one day post intervention | Assessed at baseline, one day post intervention.
  The step length will be recorded in meters.
Change from Baseline arm ROM maximum at one day post intervention | Assessed at baseline, one day post intervention.
  The arm ROM maximum will be recorded in degree.
Change from Baseline turning average duration velocity at one day post intervention | Assessed at baseline, one day post intervention.
  The turning average duration velocity will be recorded in cm/s.
Change from Baseline gait cycle at one day post intervention | Assessed at baseline, one day post intervention.
  The gait cycle will be recorded in s.
Change from Baseline Unified Parkinson's Disease Rating Scale-III at one day post intervention | Assessed at baseline, one day post intervention.
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms.
Changes in Tinetti Gait scores at one day post intervention | Assessed at baseline, one day post intervention.
  This indicator mainly reflects the stability of posture .
Changes in Tinetti Balance scores at one day post intervention | Assessed at baseline, one day post intervention.
  This indicator mainly reflects the stability of gait.

SECONDARY OUTCOMES:
Changes in ΔHbO2 concentration in the brain cortex | Assessed at baseline, one day post intervention.
  The ΔHbO2 concentration in the brain cortex will be recorded in oxyhemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Kezhong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No